CLINICAL TRIAL: NCT00849823
Title: A Brief, Clinic-Based, HIV Prevention Program for African American Teen Males
Brief Title: HIV Prevention Program for African American Teen Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Crosby (Other)
Collaborators: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor-Investigator, Richard Crosby, Chair-Department of Health Behavior, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 080666; NIH Grant # 1R01MH083621
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: HIV Infections; Sexually Transmitted Infections
Keywords: African American; Men; Condoms; Randomization; Brief Intervention; HIV; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Male Sexual Health Program (Active Comparator)
  Interventions: Behavioral: Male Sexual Health Program
- Focus on the Future Program (Experimental)
  Interventions: Behavioral: Focus on the Future Program

INTERVENTIONS:
Behavioral: Male Sexual Health Program — An attention equivalent control condition entailing a 60-minute one-to-one session that will didactically teach teens about several aspects of male sexual health. The content and objectives are related only to knowledge acquisition. In addition to this program, teens randomized to the control condition will receive standard-of-care services from the clinic. This involves the provision of free condoms (one size "fits all" condoms) and a brief (nurse-delivered) counseling message to practice safer sex.
  Arms: Male Sexual Health Program
Behavioral: Focus on the Future Program — A 60-minute, theory-guided program designed to increase the quality and frequency of teens' condom use within the context of making safer choices regarding partners and sexual behaviors. The program is explicitly designed to increase the quality and frequency of teen's condom use.
  Arms: Focus on the Future Program

SUMMARY:
The purpose of this study is to test if sexual health interventions can reduce the incidence of STIs among African American teens (15 to 21 years old). By doing this study, we hope to help African American teens improve their condom use skills and encourage them to use condoms more frequently. If the number of STIs in this population can be decreased, the health of African American teen males will greatly improve. We also believe that sexual partners (typically African American teen females) will also benefit.

DETAILED DESCRIPTION:
Based on the observation that African Americans are vastly more likely than their white and Hispanic counterparts to be infected by the human immunodeficiency virus (HIV), the Centers for Disease Control and Prevention (CDC) has termed AIDS a "health crisis" for African Americans and has called for a heightened national response to this glaring racial disparity. The crisis is especially dramatic in the Southern United States. Thus, the search for effective interventions tailored to this population is a national priority. This study expands upon a previous study conducted among young African American men. In the previous study we developed and tested the efficacy of a brief, clinic-based, program designed to interactively promote safer sex for African American men (18 to 29 years of age) engaging in sex with women. Adjusted findings from the previous study provided relatively robust support for program efficacy, with men who received the intervention program being about two-thirds less likely, than controls, to acquire an STI during a 6-month period. This study expands on the work performed in the previous study by developing and testing a version for younger African American males (i.e., teen males).

The purpose of this study is to test the efficacy of a brief, clinic-based and theory-guided, intervention designed to reduce STI incidence among African American teen (15 to 20 years old) males presenting themselves for STI testing.

ELIGIBILITY:
Inclusion Criteria:

* at least 15, but not more than 23 years of age
* attending the clinic for the expressed purpose of being tested for sexually transmitted infections
* engaging in penetrative sex (penile-vaginal or penile-anal) at least once in the past 2 months
* willingness to return for the two planned follow-up assessments

Exclusion Criteria:

* self-report of being HIV positive

Ages: 15 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 840 (Estimated)
Dates: Start 2009-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence rate of laboratory-confirmed STIs | 2- and 6-month follow-up, as well as 12-month follow-up medical records review
Self-report of unprotected penetrative sex (past 30 days) | 2- and 6-month follow-up
Self-report of number of penetrative (penile-vaginal or penile-anal) sex partners (past 30 days) | 2 and 6-month follow-up
Self-report of negative experiences with the correct use of condoms (past 30 days) | 2- and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Pasternak, MD, MPH, Principal Investigator — Louisiana State University Health Sciences Center in New Orleans; Richard A Crosby, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Adolescent Medicine Program, LSU School of Medicine, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Crosby RA, Mena L, Smith RV. Promoting positive condom use experiences among young black MSM: a randomized controlled trial of a brief, clinic-based intervention. Health Educ Res. 2018 Jun 1;33(3):197-204. doi: 10.1093/her/cyy010. PMID 29534210
- [Derived] Crosby RA, Mena L, Salazar LF, Hardin JW, Brown T, Vickers Smith R. Efficacy of a Clinic-Based Safer Sex Program for Human Immunodeficiency Virus-Uninfected and Human Immunodeficiency Virus-Infected Young Black Men Who Have Sex With Men: A Randomized Controlled Trial. Sex Transm Dis. 2018 Mar;45(3):169-176. doi: 10.1097/OLQ.0000000000000721. PMID 29419709
- [Derived] Crosby R, Salazar LF. Reduction of condom use errors from a brief, clinic-based intervention: a secondary analysis of data from a randomised, controlled trial of young black males. Sex Transm Infect. 2015 Mar;91(2):111-5. doi: 10.1136/sextrans-2013-051492. Epub 2014 Jun 4. PMID 24898858